CLINICAL TRIAL: NCT03639636
Title: Comparative Evaluation of Serum Sclerostin in Chronic Periodontitis Patients Before and After Surgical Periodontal Therapy in Conjunction With Nonsurgical Periodontal Therapy
Brief Title: is the Sclerostin Marker of Chronic Periodontitis
Acronym: itsmcp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Banda Madhavi, Dr.banda madhavi, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: madhavisclerostin
Record Dates: First submitted 2018-08-10; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Periodontitis
Keywords: periodontitis; sclerostin; periodontal surgery; scaling and root planing
MeSH Terms: conditions — Periodontitis; Sclerosteosis

STUDY DESIGN:
Intervention Model Description: interventional prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional prospective study (Other): nonsurgical periodontal therapy(scaling and root planing) surgical therapy( flap surgery)
  Interventions: Other: non surgical and surgical periodontal therapy

INTERVENTIONS:
Other: non surgical and surgical periodontal therapy — scaling and root planing periodontal flap surgery

SUMMARY:
Reviewed literature suggests that sclerostin will inhibit the bone formation and ultimately leads to chronic periodontitis. Estimation of Sclerostin levels in the serum of periodontitis patients before and after intervention could explore the effectiveness of therapy and also give a more detailed insight into its diagnostic and prognostic potential as a biomarker of periodontal disease.

DETAILED DESCRIPTION:
Advances during the last decade provided relevant information on the regulation of Sost/sclerostin and its mechanism(s) of action. Several stimuli have been reported to regulate Sost/Sclerostin expression, however how these factors interplay to regulate the expression of this gene in a spatiotemporal manner is unknown. Animal studies demonstrate that sclerostin is key for skeletal homeostasis, and required for the bone anabolic response to mechanical loading although appears dispensable for PTH-induced bone gain. The knowledge provided by preclinical investigations resulted in clinical trials based on the neutralization of sclerostin activity as a novel osteoanabolic therapeutic approach. It is now clear that sclerostin is capable of uncoupling bone formation and bone resorption, by inhibiting osteoblast function while stimulating osteoclast function, as the bone gain achieved by pharmacologic inhibition of sclerostin results from stimulation of osteoblast activity and inhibition of bone resorption. Furthermore, the recent observations show that activation of βcatenin in osteocytes increases bone resorption and Rankl production in a sclerostin-dependent manner. Anti-sclerostin therapy has shown beneficial skeletal outcomes in osteoporotic patients, however more recent evidence shows that the anabolic effects of this therapy attenuate with time and that after discontinuation BMD returns to pretreatment levels over time. The new evidence showing increased levels of Sost/sclerostin (and Dkk1) after activation of Wnt-βcatenin signaling suggest that sclerostin (and Dkk1) act as a negative feedback limiting bone formation stimulated by this pathway.

In this study is there any alterations in sclerostin levels in serum response to periodontal therapy was checked. Periodontal therapy alters the inflammation pathway is a proven fact.

ELIGIBILITY:
Inclusion Criteria:• Systemically healthy individuals with more than 50% remaining natural teeth

* All the patients who are diagnosed as having generalized chronic periodontitis based on the American Academy of Periodontology (AAP) classification.
* Probing Pocket Depth (PPD)/ Clinical Attachment Loss(CAL) ≥ 5mm
* Patients indicated for periodontal surgery

Exclusion Criteria:• The patients who have aggressive periodontitis/localized periodontitis

* Patients having any other systemic diseases
* Patients taking high-dose steroid therapy, radiation or immunosuppressive therapy and any other drug history.
* Pregnant and lactating woman.
* History of smoking within the past five years.
* Patients who had undergone periodontal therapy in the last six months.
* Intellectual disability

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
sclerostin level response to only scaling and root planing | 4 weeks
  measuring serum sclerostin levels in pg/ml(Pico grams per milli liter),

SECONDARY OUTCOMES:
sclerostin level response to periodontal surgery | 6 weeks
  measuring serum sclerostin levels after surgery in pg/ml(Pico grams per milli liter)

OTHER OUTCOMES:
periodontal parametors | 0-4-6 weeks
  pocket probing depth,Clinical Attachment Level(CAL), both are in mm

CONTACTS AND LOCATIONS:
Overall Officials: Jammula surya prasanna, mds, Study Director — panineeya institute of dental sciences and research center
Locations (1):
- Panineeya Institute of Dentalsciences and Research Center, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu M, Kurimoto P, Zhang J, Niu QT, Stolina M, Dechow PC, Feng JQ, Hesterman J, Silva MD, Ominsky MS, Richards WG, Ke H, Kostenuik PJ. Sclerostin and DKK1 Inhibition Preserves and Augments Alveolar Bone Volume and Architecture in Rats with Alveolar Bone Loss. J Dent Res. 2018 Aug;97(9):1031-1038. doi: 10.1177/0022034518766874. Epub 2018 Apr 4. PMID 29617179
- [Background] Chen H, Xu X, Liu M, Zhang W, Ke HZ, Qin A, Tang T, Lu E. Sclerostin antibody treatment causes greater alveolar crest height and bone mass in an ovariectomized rat model of localized periodontitis. Bone. 2015 Jul;76:141-8. doi: 10.1016/j.bone.2015.04.002. Epub 2015 Apr 11. PMID 25868799
- [Result] Taut AD, Jin Q, Chung JH, Galindo-Moreno P, Yi ES, Sugai JV, Ke HZ, Liu M, Giannobile WV. Sclerostin antibody stimulates bone regeneration after experimental periodontitis. J Bone Miner Res. 2013 Nov;28(11):2347-56. doi: 10.1002/jbmr.1984. PMID 23712325
- [Result] Balli U, Aydogdu A, Dede FO, Turer CC, Guven B. Gingival Crevicular Fluid Levels of Sclerostin, Osteoprotegerin, and Receptor Activator of Nuclear Factor-kappaB Ligand in Periodontitis. J Periodontol. 2015 Dec;86(12):1396-404. doi: 10.1902/jop.2015.150270. Epub 2015 Sep 14. PMID 26367496